CLINICAL TRIAL: NCT03885635
Title: Hemiarch vs Extended Arch in Aortic Dissection - a SystemaTic Analysis by Randomized Trial (HEADSTART)
Brief Title: Hemiarch vs Extended Arch in Type 1 Aortic Dissection
Acronym: HEADSTART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEADSTART
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Intervention Model Description: Hemiarch vs. extended arch repair in the setting of acute DeBakey type 1 aortic dissections
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemiarch repair (Active Comparator): Standard hemiarch repair with open distal anastomosis in the proximal arch without replacement of the head vessels.
  Interventions: Procedure: Hemiarch repair
- Extended arch repair (Active Comparator): Ascending aortic and arch replacement with or without head vessel re-implantation and single TEVAR device placement within 1 week.
  Interventions: Procedure: Extended arch repair

INTERVENTIONS:
Procedure: Hemiarch repair — Current standard of surgical repair consisting of ascending aortic replacement with open distal anastomosis at level of proximal arch under a period of hypothermic circulatory arrest . No surgical or endovascular intervention is carried out in the mid arch or descending aorta. Intra-operative management, including cannulation, cardioplegia, cerebral perfusion technique, and neurologic monitoring will be done according to each institution's current standard of practice.
  Arms: Hemiarch repair
Procedure: Extended arch repair — Surgical replacement of the ascending aorta along with intervention on the arch and descending aorta. Techniques for distal aspect of extended arch technique include but are not limited to total arch replacement along with TEVAR, Frozen Elephant Trunk procedure or surgical proximal arch replacement with bare metal stents in arch and descending aorta. Intra-operative management, including cannulation, cardioplegia, cerebral perfusion technique, and neurologic monitoring will be done according to each institution's current standard of practice.
  Arms: Extended arch repair

SUMMARY:
HEADSTART is a prospective, open-label, non-blinded, multicenter, randomized controlled trial that compares a composite of mortality and re-intervention in patients undergoing hemiarch and extended arch repair for acute DeBakey type 1 aortic dissection. Eligible patients will be randomized to one or the other surgical strategy and clinical and imaging outcome data will be collected over a 3 year follow up period.

DETAILED DESCRIPTION:
DeBakey Type 1 aortic dissections continue to have high operative mortality and morbidity and there is equipoise in available literature with regards to the best operative strategy and patient selection criteria. Hemiarch repair is current standard of care in most centers but extended arch repair is gaining popularity aiming to address early post-operative malperfusion and improve long term aortic remodeling.

HEADSTART is a randomized controlled prospective trial of patients presenting to participating institutes with acute DeBakey 1 aortic dissection. Patients will be enrolled and randomized into one of two groups - 'hemiarch repair' and 'extended arch repair'. Pre-operative, early post-operative and long term follow clinical and CT imaging data will be collated on a centralized database and at a core lab respectively.

ELIGIBILITY:
Inclusion Criteria

1. Emergent surgical repair of Acute DeBakey Type 1 aortic dissection
2. Age >18 years and <70 years
3. Operating surgeon believes that both surgeries could be safe and effective

Exclusion Criteria

1. Hemodynamic instability/shock defined as systolic BP < 90 mm Hg
2. Previous cardiac surgery with sternotomy or thoracic endograft placement
3. Aortic arch diameter > 6cm in which a concomitant arch replacement is judged necessary
4. Procedures deemed to be "salvage operations" where the patient is unlikely to survive hospital discharge.
5. GCS < 8 for more than 6 hours
6. History of cirrhosis.
7. History of chronic renal failure (baseline eGFR < 50)
8. Metastatic malignancy
9. Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing a composite end-point of mortality or re-intervention | 3 years
  Compare the proportion of patients between the two groups who over a 3 year follow up period attain a composite clinical end-point of 1) mortality, 2) late aortic re-intervention, either surgical or endovascular (> 30 days from index procedure) or 3) early (< 30 days from index procedure) re-intervention for branch malperfusion

SECONDARY OUTCOMES:
Number of patients achieving complete false lumen thrombosis on CT imaging | 3 years
  Compare the proportions of patients achieving complete false lumen (FL) thrombosis in the proximal, mid and distal descending thoracic aorta at 3 years after intervention between the two groups
Delta change in the ratio of true lumen to total aortic area (TL: Ao) | 1 month
  Compare delta change in the ratio of true lumen to total aortic area (TL:Ao) in the descending thoracic and abdominal aorta from pre-operative to first post-operative CT scans, between the two groups.
Delta change in maximum cross-sectional descending thoracic aortic dimension | 3 years
  Compare delta change in the maximum cross-sectional descending thoracic dimension between the two groups over 3 years
Number of patients experiencing the listed peri-operative complications | 1 month
  To compare the proportion of patients experiencing the following peri-operative complications between the two groups: mortality, stroke, paraplegia/paraparesis, vascular injury, renal ischemia, bowel ischemia warranting operative intervention, peripheral limb ischemic changes and re-operation for bleeding.
Number of patients requiring open surgical or endovascular re-intervention | 3 years
  Compare the proportion of patients requiring open surgical and endovascular re-intervention over 3 years in both groups
Preoperative malperfusion and perioperative mortality/early re-intervention | 1 month
  Correlate pre-operative CT signs of malperfusion with peri-operative mortality and early post-operative re-intervention in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Munir Boodhwani, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Jehangir Appoo, MD, Principal Investigator — University of Calgary
Locations (4):
- Canada (4):
  - London Health Sciences Centre, London, Ontario
  - University Health Network, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire De Cardiologie Et De Pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elbatarny M, Stevens LM, Dagenais F, Peterson MD, Vervoort D, El-Hamamsy I, Moon M, Al-Atassi T, Chung J, Boodhwani M, Chu MWA, Ouzounian M; Canadian Thoracic Aortic Collaborative Investigators. Hemiarch versus extended arch repair for acute type A dissection: Results from a multicenter national registry. J Thorac Cardiovasc Surg. 2024 Mar;167(3):935-943.e5. doi: 10.1016/j.jtcvs.2023.04.012. Epub 2023 Apr 20. PMID 37084820